CLINICAL TRIAL: NCT04301440
Title: THE PHYSIOLOGICAL EFFECTS OF ELECTROMAGNETIC EMISSIONS ON THE GENERAL CONDITION OF THE PATIENT
Acronym: EPHEME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Bizet (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-A03150-57
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Electromagnetic Emissions and Emotional Disorder; Electromagnetic Emissions and Medication Savings
Keywords: Anxiety; Depression; Quality of life; Medication savings; Electromagnetic emissions
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The study concerns adult patients hospitalized for the management of a chronic pathology and / or its complications
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with anxious and / or depressive characteristics : treated group (Active Comparator): patients with anxious and / or depressive characteristics, The device with the electromagnetic wave will be connected
  Interventions: Device: The emission of electromagnetic with the probes
- patients with anxious and / or depressive characteristics : placebo group (Placebo Comparator): The device with the electromagnetic wave will not be connected
  Interventions: Device: The emission of electromagnetic without the probes

INTERVENTIONS:
Device: The emission of electromagnetic with the probes — The patient will be in the lying position, a probe will be positioned in the middle of the chest and the second probe below the xyphoid. The probes will be fixed by a band to keep them in place. The emission of electromagnetic waves is painless.
  Arms: patients with anxious and / or depressive characteristics : treated group
Device: The emission of electromagnetic without the probes — The patient will be in the lying position, a probe will be positioned in the middle of the chest and the second probe below the xyphoid. The probes will be fixed by a band to keep them in place. The emission of electromagnetic waves is painless.
  Arms: patients with anxious and / or depressive characteristics : placebo group

SUMMARY:
Hospital patients usually experience anxiety caused by physiological, psychological and environmental stimuli. This emotional state corresponds to the psychophysiological response to a perceived threat.

The investigator's goal is to use a non-drug approach to these problems which would help improve the quality of life of patients, prevent the consumption of anti-anxiety drugs / antidepressants; and thus to reduce the direct cost in terms of treatment, but also to reduce the indirect costs linked to work stoppages and the consumption of the care offer.

Working hypothesis: Local magnetic muscle stimulation improves people's well-being and relaxation

DETAILED DESCRIPTION:
Primary objective :

Describe the effect of the intervention on the level of anxiety / depression in patients with anxious and / or depressive characteristics

Secondary objectives:

* Describe the variation in the quality of life of patients before and after the intervention
* Describe the variation in drug consumption
* Describe the use of post intervention hospitalization
* Describe the variation in the quality of sleep before and after the intervention
* Describe the timeframe for returning patients to professional activity

ELIGIBILITY:
Inclusion Criteria:

* Major patient hospitalized for the management of a chronic pathology and / or its complications;
* Patient with a Hospital Anxiety and Depression scale score (HAD) ≥ 8 for items assessing anxiety disorders; AND a HAD score ≥ 8 for the items assessing depressive disorders.
* Subject affiliated to a social security scheme or beneficiary of such a scheme
* No participation in another clinical study

Exclusion Criteria:

* Minor patient
* Pregnant and breastfeeding women
* HAD score <8 for items evaluating anxiety disorders OR a HAD score <8 for items evaluating depressive disorders
* Major subject protected by law, under curatorship or tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Improved quality of life in depressed and anxiety patients: Hospital Anxiety and Depression scale | Ten days
  Evaluation with Hospital Anxiety and Depression scale
Decreased consumption of anti-anxiety and anti-depressant drugs | Ten days
  Prescription analysis
Improved quality of sleep: Epworth scale | Ten days
  Evaluation with Epworth scale

CONTACTS AND LOCATIONS:
Locations (1):
- Benkessou, Paris, France